CLINICAL TRIAL: NCT05103644
Title: Study of the Therapeutic Effect of Atorvastatin on the Clinical Outcomes in HER2 Negative Breast Cancer Patients"
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, ALshaimaa Ibrahim Rabie, clinical pharmacist Msc, Pharm D, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMBSUREC/10102021/Rabie
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: study group control group
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): breast cancer patient received Atorvastatin 80 mg
  Interventions: Drug: Atorvastatin 80mg
- control group (Placebo Comparator): breast cancer patient received placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Atorvastatin 80mg — patients received statin experimental group
  Other Names: ATOR
  Arms: study
Other: placebo — patients received placebo control group
  Other Names: placebo single blind
  Arms: control group

SUMMARY:
Statins, a major class of drugs for treatment of hypercholesterolemia, are widely used due to a notable prevention of cardiovascular disease, and accumulating evidence proposes a promising role of statins in breast cancer

DETAILED DESCRIPTION:
Statin has lipid independent effects include inhibition of inflammatory responses, immunomodulatory actions, apoptotic and antiproliferative effects, which might contribute to the suggested anti-tumoral effects of these agents. The epidemiological evidence projecting statins as anticancer agents is variable, depending on the particular type of cancer in question as well as the class of statin used

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed breast cancer any stage confirmed by radiological and pathological or by clinical evaluation undergo surgery or receiving neo/adjuvant chemotherapy treatment
2. Age above 18 years
3. HER2 negative core biopsy
4. Adequate renal function: the calculated creatinine clearance should be ≥50 mL/min
5. Patients must be accessible for treatment and follow-up
6. Performance status of Eastern Cooperative Oncology Group (ECOG) ≤ 2

Exclusion Criteria:

1. Known hypersensitivity reaction to the investigational compounds or incorporated substances
2. patients who are unlikely to comply with trial requirements (eg, confusion, psychological or mood disturbances ,alcoholism, cardiac arrhythmia)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Femal breast cancer
Enrollment: 60 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Ki-67 molecular | 3 month
  antiproliferative effect Ki-67 molecular gene expression
TAZ (WWTR1) TAZ expression | 3 months
  cell proliferative ability via TAZ (WWTR1) TAZ expression
cardiac markers | 3 months
  protective effect of atorvastatin for Anthracycline induced cardiotoxicity

SECONDARY OUTCOMES:
Overall survival OS | time frame 6 month
  The length of time from r the start of treatment for a disease and are still alive
Overall response rate | 6 months
  the proportion of patients who have a partial or complete response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hassan shaaban, MD, Study Director — Beni-Suef University; Raghda RS Hussein, PHD, Study Director — Beni-Suef University; Reham shehab El-Nemr, MD, Study Director — Fayoum University
Locations (2):
- Egypt (2):
  - Fayoum Oncology Center, Al Fayyum
  - Beni-Suef university hospital, Banī Suwayf